CLINICAL TRIAL: NCT01959503
Title: A Prospective, Randomized Study to Compare Progel Vascular Sealant to Gelfoam Plus as an Adjunct for the Control of Bleeding in Subjects Undergoing Thoracic Aortic Surgery
Brief Title: Progel Vascular Sealant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEO13-100
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Aortic Valve Stenosis; Aneurysm of Ascending Aorta; Aortic Valve Disorder; Bicuspid Valve Disorder
Keywords: Aorta; Aortic; Reconstruction; CABG; Bypass
MeSH Terms: conditions — Aortic Valve Stenosis; Aneurysm, Ascending Aorta; Aortic Valve Disease | interventions — Gelatin Sponge, Absorbable

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Progel Vascular Sealant (Experimental): Progel Vascular Sealant after confirmation of anastomotic leakage during intra-procedure leak test.
  Interventions: Device: Progel Vascular Sealant
- Gelfoam Plus (Active Comparator): Gelfoam Plus Sealant after confirmation of anastomotic leakage during intra-procedure leak test.
  Interventions: Device: Gelfoam Plus

INTERVENTIONS:
Device: Progel Vascular Sealant
  Other Names: Progel
  Arms: Progel Vascular Sealant
Device: Gelfoam Plus
  Other Names: Gelfoam
  Arms: Gelfoam Plus

SUMMARY:
This study is being conducted to evaluate the safety and effectiveness of the Progel Vascular Sealant for use in vascular reconstructions to achieve adjunctive hemostasis by mechanically sealing areas of leakage.

DETAILED DESCRIPTION:
The primary objective of this clinical study is to compare the time to hemostasis at the aortic anastomotic suture line in subjects receiving Progel (Test group) to that in subjects receiving Gelfoam Plus (Control group) on anastomotic suture lines involving the aortic valve, ascending aorta, or aortic arch while on cardiopulmonary bypass.

The primary endpoint of this study is the time to achieve hemostasis at the aortic anastomotic suture line from the time surgical clamps are released to cessation of leakage at the treated anastomotic site with either Progel (Test) or Gelfoam Plus (Control).

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject must be ≥ 18 years of age.
* 2. Subject is scheduled for elective, primary thoracic surgery involving the aortic valve, ascending aorta, or aortic arch on cardiopulmonary bypass.
* 3. Subject has an expected life expectancy> 6 months.
* 4. Subject is willing and able to comply with all aspects of the study including follow-up schedule.
* 5. Subject or authorized representative, has the ability to provide voluntary written informed consent.

Intra-operative Inclusion Criteria:

* 1. Subject is able to undergo an antegrade cardioplegia injection for evaluation of a leak at the aortic anastomotic site(s) during the procedure.
* 2. Following this injection, subject has a leaking site where a topical sealant/hemostatic agent may be used to control bleeding.

Exclusion Criteria:

* 1. Subject has Type A or other acute thoracic aortic dissection.
* 2. Subject has undergone prior thoracic surgery (open thoracotomy not including interventional cardiology procedures).
* 3. Subject is undergoing a planned concomitant procedure other than coronary artery bypass graft (CABG).
* 4. Subject has a previous organ transplant.
* 5. Subject has known or suspected preoperative coagulation disorder.
* 6. Subject is allergic to human thrombin or has a history of allergic reactions after application of human thrombin.
* 7. Subject is allergic to protamine.
* 8. Subject has a Left Ventricular Assist Device (LVAD) or planned to receive an LVAD.
* 9. Subject is undergoing emergency surgery.
* 10. Subject is in chronic renal failure.
* 11. Subject has a hematocrit < 21% pre-operatively.
* 12. Subject has a serum creatinine ≥2.5 mg/dl at baseline or is currently on dialysis.
* 13. Subject has a cardiac ejection fraction <25%.
* 14. Subject is scheduled for another cardiac surgery within 30 days of enrollment.
* 15. Subject has an active or latent infection which is systemic or at the intended surgery site.
* 16. Subject is immuno-compromised such as that resulting from chronic oral steroid use, chemotherapeutic agents, or immune deficiency disorders.
* 17. Subject is pregnant by a positive pregnancy test or has plans to become pregnant during the study period or is currently breast-feeding.
* 18. Subject is unwilling to receive blood products.
* 19. Subject has participated in another investigational research study within 30 days of enrollment.
* 20. In the opinion of the investigator, the subject has a clinical condition that would preclude the use of the study device, preclude the subject from completing the follow-up requirements, or would complicate the evaluation of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Khoynezhad, MD, Principal Investigator — Cedars-Sinai Heart Institute
Locations (19):
- United States (19):
  - Cedars-Sinai, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Portneuf Hospital, Pocatello, Idaho
  - Northwestern University, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Hospital, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Bryan Heart, Lincoln, Nebraska
  - Cornell University, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolinas Health Care System, Charlotte, North Carolina
  - Ohio Health Research Institute, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Houston Methodist Hospital, Houston, Texas
  - The Heart Hospital Baylor, Plano, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia Health Sciences Center, Charlottesville, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia

REFERENCES:
- [Derived] Ma GW, Kucey A, Tyagi SC, Papia G, Kucey DS, Varcoe RL, Forbes T, Neville R, Dueck AD, Kayssi A. The role of sealants for achieving anastomotic hemostasis in vascular surgery. Cochrane Database Syst Rev. 2024 May 2;5(5):CD013421. doi: 10.1002/14651858.CD013421.pub2. PMID 38695613

RESULTS

PARTICIPANT FLOW:
Groups:
- Progel Vascular Sealant: Progel Vascular Sealant after confirmation of anastomotic leakage during intra-procedure leak test.
  Progel Vascular Sealant
- Gelfoam Plus: Gelfoam Plus Sealant after confirmation of anastomotic leakage during intra-procedure leak test.
  Gelfoam Plus
Period: Overall Study
Arm/Group | Progel Vascular Sealant | Gelfoam Plus
Started | 107 | 51
Completed | 104 | 49
Not Completed | 3 | 2
Not completed — Death | 2 | 1
Not completed — Randomized but not treated | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants who were randomized and treated
Groups:
- Total: Total of all reporting groups
Arm/Group | Progel Vascular Sealant | Gelfoam Plus | Total
Number analyzed (Participants) | 106 | 50 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (14.42) | 62.4 (14.30) | 61.8 (14.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 15 | 47
  Male | 74 | 35 | 109
Region of Enrollment [Number; unit: participants]
  United States | 106 | 50 | 156

OUTCOME MEASURES:

1. Primary Outcome: Time to Achieve Hemostasis at the Aortic Anastomotic Suture Line From the Time Surgical Clamps Are Released to Cessation of Leakage at the Treated Anastomotic Site With Either Progel or Gelfoam.
Time Frame: 0 seconds to 600 seconds
Population: In the Progel group one subject was not evaluable as information was not collected for the primary end-point changing the number from 106 to 105, compare to baseline characteristics.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Progel Vascular Sealant | Gelfoam Plus
Number analyzed (Participants) | 105 | 50
seconds | 124.3 (202.09) | 377.8 (252.4)
Statistical Analysis 1: Comparison: Progel Vascular Sealant vs Gelfoam Plus; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank-Sum Test

2. Secondary Outcome: Proportion of Subjects Who Achieve Successful Hemostasis at All Treated Aortic Anastomotic Suture Lines Following Assigned Treatment.
Time Frame: 5 minutes after application
Population: In the Progel group one subject was not evaluable as information was not collected for this endpoint, which change the number from 106 to 105, compare to baseline characteristics.
Measure: Number; unit: percentage of participants
Arm/Group | Progel Vascular Sealant | Gelfoam Plus
Number analyzed (Participants) | 105 | 50
percentage of participants | 85.7 | 40.0
Statistical Analysis 1: Comparison: Progel Vascular Sealant vs Gelfoam Plus; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 9.00, 95% CI 2-sided [4.07 to 19.89]

3. Secondary Outcome: Proportion of Subjects Who Achieve Immediate Hemostasis, Defined as 0 Seconds, at All Treated Aortic Anastomotic Suture Lines Following Assigned Treatment.
Time Frame: 0 seconds to 10 minutes
Measure: Number; unit: percentage of participants
Arm/Group | Progel Vascular Sealant | Gelfoam Plus
Number analyzed (Participants) | 106 | 50
percentage of participants | 59.4 | 16.0
Statistical Analysis 1: Comparison: Progel Vascular Sealant vs Gelfoam Plus; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 7.69, 95% CI 2-sided [3.27 to 18.11]

4. Secondary Outcome: Chest Tube Drainage Volume Following Surgery.
Time Frame: 24 hours post procedure
Population: In the Gelfoam Plus group one subject was not evaluable as information was not collected for this endpoint, which change the number from 50 to 49, compare to baseline characteristics.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Progel Vascular Sealant | Gelfoam Plus
Number analyzed (Participants) | 106 | 49
mL | 701.6 (499.83) | 589.6 (359.41)

5. Secondary Outcome: Proportion of Subjects Who Received Transfusion Within 24 Hours Following Surgery
Time Frame: 24 hours post procedure
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Progel Vascular Sealant | Gelfoam Plus
Number analyzed (Participants) | 106 | 49
participants | 46 | 19

6. Secondary Outcome: Time Between Cross Clamp Removal and Request of Surgical Wires for Sternal Closure.
Time Frame: Intra-procedurally
Population: In the Vascular group two subjects were not evaluable as information was not collected for this endpoint, which changes the number from 106 to 104, compare to baseline characteristics.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Progel Vascular Sealant | Gelfoam Plus
Number analyzed (Participants) | 104 | 50
minutes | 59.4 (30.96) | 58.5 (24.74)

7. Secondary Outcome: Incidence of Reoperations for Aortic Bleeding Complications Following Treatment.
Time Frame: 30 days post procedure
Measure: Number; unit: participants
Arm/Group | Progel Vascular Sealant | Gelfoam Plus
Number analyzed (Participants) | 106 | 50
participants | 0 | 1

8. Secondary Outcome: Proportion of Subjects With Device-Related Serious Adverse Events Following Assigned Treatment Through 30 Days
Time Frame: 30 days post procedure
Population: One subject in Progel Vascular Sealant and one subject in Gelfoam Plus discontinue before 30days and do not have device-related SAE. They are considered as not evaluable and are not included in this analysis, thus makes the difference compared to population in baseline.
Measure: Number; unit: participants
Arm/Group | Progel Vascular Sealant | Gelfoam Plus
Number analyzed (Participants) | 105 | 49
participants | 3 | 4

ADVERSE EVENTS:
Time Frame: Incidence of reoperations for aortic bleeding complications following assigned treatment through 30 days. Number of device-related serious adverse events per patient following assigned treatment through 30 days.
Arm/Group | Progel Vascular Sealant | Gelfoam Plus
Serious Adverse Events (participants affected / at risk) | 51/106 | 29/50
Other Adverse Events (participants affected / at risk) | 51/106 | 29/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Progel Vascular Sealant (N=106) | Gelfoam Plus (N=50)
Anemia (Blood and lymphatic system disorders) | 5 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 27 | 17
Atrial flutter (Cardiac disorders) | 2 | 3
Atrioventricular block (Cardiac disorders) | 2 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 2
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 2 | 0
Cardiogenic shock (Cardiac disorders) | 2 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Ischemic cardiomyopathy (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Pericardial hemorrhage (Cardiac disorders) | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 2
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Melena (Gastrointestinal disorders) | 1 | 0
Complication of device removal (General disorders) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Incision site infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 | 0
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 2 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 2
Convulsion (Nervous system disorders) | 0 | 1
Embolic stroke (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Renal injury (Renal and urinary disorders) | 2 | 0
Renal tubular acidosis (Renal and urinary disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Mediastinal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Incisional drainage (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hematoma (Vascular disorders) | 1 | 1
Hemorrhage (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Hypovolemic shock (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Progel Vascular Sealant (N=106) | Gelfoam Plus (N=50)
Anemia (Blood and lymphatic system disorders) | 34 | 12
Leukocytosis (Blood and lymphatic system disorders) | 25 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 19 | 7
Atrial Fibrillation (Cardiac disorders) | 13 | 7
Tachycardia (Cardiac disorders) | 6 | 2
Nausea (Gastrointestinal disorders) | 15 | 7
Vomiting (Gastrointestinal disorders) | 1 | 4
Fatigue (General disorders) | 3 | 5
Oedema Peripheral (General disorders) | 18 | 4
Pyrexia (General disorders) | 2 | 3
Fluid Overload (Metabolism and nutrition disorders) | 10 | 8
Hyperglycemia (Metabolism and nutrition disorders) | 8 | 5
Hypokalemia (Metabolism and nutrition disorders) | 7 | 2
Hyponatremia (Metabolism and nutrition disorders) | 3 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 7 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Dizziness (Nervous system disorders) | 6 | 3
Renal Injury (Renal and urinary disorders) | 5 | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 36 | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 38 | 17
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 10 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Hypotension (Vascular disorders) | 13 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
INSTITUTION and INVESTIGATOR agree if the Study is part of a multi-center study, the first publication of the results of the Study shall be made in coajunction with the results from the investigators at the other Study centers. In the event no publication of the multi-center study has been made within two years after the completion of the Study at all Study centers, then INSTITUTION and INVESTIGATOR shall be free to publish the Study results generated.